CLINICAL TRIAL: NCT02410681
Title: Associations Between Sleep Bruxism and (Peri-)Implant Complications: a Follow-up Study
Brief Title: Sleep Bruxism and (Peri-)Implant Complications
Status: Completed | Type: Observational
Sponsor: Frank Lobbezoo (Other)
Responsible Party: Sponsor-Investigator, Frank Lobbezoo, Prof. Dr., Academic Centre for Dentistry in Amsterdam
Organization: Academic Centre for Dentistry in Amsterdam (Other)
Other Study IDs: ACTA_2012-2015
Record Dates: First submitted 2015-03-26; First posted 2015-04-08 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Dental Implant Complications; Sleep Bruxism
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peri-implant intrasulcular biofilm.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Electromyographic recording of temporalis muscle activity during sleep — Electromyographic recording of temporalis muscle activity during sleep. In total, 9 sleep recordings will be done at the home setting of each participant.
  1. 3 recordings after the baseline visit
  2. 3 recordings 6 weeks after the baseline visit
  3. 3 recordings one year after the baseline visit
Radiation: Vertical bitewing radiograph — An intraoral vertical bitewing radiograph will be performed with the assistance of individually modified plate positioning devices at each visit (in total 8 visits during the 2-year follow-up period).
Other: Collection of biofilm sample — Collection of peri-implant intrasulcular biofilm sample for DNA analysis of the biofilm composition. In total, samples will be collected three times:
  1. At the baseline visit
  2. Three months after the baseline visit
  3. One year after the baseline visit

SUMMARY:
Excessive mechanical forces can cause complications of dental implants and their suprastructures (crowns and bridges), and can possibly be destructive for the bone and soft tissues around the implants. Sleep bruxism (grinding and clenching of the teeth during sleep) is considered as an important source of mechanical forces in the oral environment. Therefore, in this study, the investigators will investigate whether sleep bruxism is associated with implant and peri-implant complications.

ELIGIBILITY:
Inclusion Criteria:

* Planned for treatment with implant-supported fixed suprastructure(s).
* 18 years of age or older.

Exclusion Criteria:

* Opposing teeth of implant-supported fixed suprastructure(s) are restored with removable artificial teeth.
* Patients categorized in the classes 3 or higher according to the ASA system for classification of physical status.
* Use of occlusal splint, mandibular repositioning appliance or any other bruxism mitigating device during sleep.
* Active periodontitis at the time of implant placement.
* Known allergy to Grindcare® electrode material.
* Patients with a pacemaker.
* Swollen, infected or inflamed tissues or skin eruptions, e.g. phlebitis, varicose veins etc. in the placement area of the Grindcare® electrode.
* Pregnant women will not be treated with dental implants. Pregnancy after placement of implants will not be a reason to stop participation of the subject in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with implant-supported fixed suprastructure(s), age 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-03; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Progression of peri-implant marginal bone loss (in mm) during a two-year follow-up period, assessed by intraoral radiographs. | Baseline, two weeks, six weeks, three months, one year, two years.
Changes in the modified Gingival Index during a two-year follow-up period, assessed by probing. | Baseline, two weeks, six weeks, three months, one year, two years.
Changes in the peri-implant clinical pocket depth (in mm) during a two-year follow-up period, assessed by probing. | Baseline, two weeks, six weeks, three months, one year, two years.
Changes in implant mobility (mobility present or not) during a two-year follow-up period, assessed by clinical examination. | Baseline, two weeks, six weeks, three months, one year, two years.
Occurrence and type of implant technical complications, assessed by clinical examination. | Six weeks, three months, one year, two years.
Changes in the peri-implant attachment level (in mm) during a two-year follow-up period, assessed by probing. | Baseline, two weeks, six weeks, three months, one year, two years.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lobbezoo, Prof. Dr., Principal Investigator — Academic Centre for Dentistry Amsterdam (ACTA)
Locations (1):
- Academic Centre for Dentistry Amsterdam (ACTA), Amsterdam, Netherlands